CLINICAL TRIAL: NCT06379568
Title: Risk of Aspergillus Infection in Patients With Chronic Structural Lung Disease
Brief Title: Risk of Aspergillus Infection in Patients With Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: SichuanPPHLC01
Record Dates: First submitted 2024-04-14; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Fungal Infection Lungs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Collect patient's blood to detect aspergillus specific IgG antibody, IgM antibody and so on
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspergillus pneumonia group: According to diagnostic criteria , patients diagnosed with IPA and CPA and were assigned to the Aspergillosis pneumonia group
  Interventions: Other: No intervention
- control group: The remaining patients without IPA and CPA were included in the Aspergillus colonization group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Large doses of systemic corticosteroids ，severe lung tissue damage and longer COPD diagnosis may increase the risk of IPA in patients with chronic structural lung disease. By comparing the risk factors of aspergillus colonization group and aspergillus infection group, the main risk factors of aspergillus pneumonia were determined.

DETAILED DESCRIPTION:
Patients with chronic lung disease were identified as positive for Aspergillus fumigatus through sputum microscopy. According to diagnostic criteria, patients diagnosed with IPA and CPA and were assigned to the Aspergillosis pneumonia group, while the remaining patients were included in the Aspergillus colonization group. Then,Risk factors for aspergillus pneumonia, invasive pulmonary aspergillus disease, and chronic pulmonary aspergillus disease, such as the use of high-dose corticosteroids, inhaled corticosteroids, and the extent of damage to basic lung structures, were identified by comparing the aspergillus colonization group with the aspergillus infection group.

ELIGIBILITY:
Inclusion Criteria:

1. Age : at least 18 years old ;
2. Imageological examination : Patients who complete high-resolution computed tomography (HRCT) images of the chest;
3. Serological examination : Patients who complete serological test results, including serum aspergillus specific IgG antibody, serum aspergillus IgM antibody and GM antigen detection.

Exclusion Criteria:

1. immunodeficiency conditions : Patients diagnosed with HIV infection, hematological malignancies, and autoimmune diseases.
2. Critically ill patients : Those who require mechanical ventilation in the ICU and have established various types of cardiopulmonary bypass.
3. Inadequate Clinical Data: Inability to provide reliable diagnostic measurements or insufficient clinical information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-repeat patients with chronic lung disease were included in the suspected pulmonary aspergillosis study group. According to the current study inclusion criteria, patients were excluded due to unqualified sputum specimens or negative culture results, together with patients lacked HRCT image data. Qualified patients were finally included. According to different group definitions, patients without IPA and CPA were classified into the Aspergillus colonization group and patients with IPA and CPA were included in the aspergillus infection group.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Descriptive statistical index | Information was collected on the day of admission
  Summarize participant characteristics using means and standard deviations for continuous variables and frequencies for categorical variables
Independent risk factor for aspergillus pneumonia | Statistical analysis was carried out after data collection within one month
  Independent risk factors for aspergillus infection were determined by multivariate logistic regression analysis.
The area under ROC curve of risk factors for aspergillus pneumonia | Statistical analysis was carried out after data collection within two month
  The area under ROC curve (AUC) was used to evaluate the classification effect of the binary classification model among Aspergillus pneumonia group, IPA group and CPA group

SECONDARY OUTCOMES:
Threshold analysis of aspergillus pneumonia | Statistical analysis was carried out after data collection within two month
  Specific cut-off values for Aspergillus specific IgG antibody × lung structural injury image score was determined to maximize diagnostic accuracy, focusing on sensitivity, specificity, and Youden index.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, doctor, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang R, Yang L, Fang H, Xie Q, Tang H, Chen L. Non-invasive monitoring of Aspergillus infections in chronic lung disease patients: a combined serology and HRCT imaging approach. Front Cell Infect Microbiol. 2025 Jun 27;15:1494522. doi: 10.3389/fcimb.2025.1494522. eCollection 2025. PMID 40654578

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT06379568/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT06379568/ICF_001.pdf